CLINICAL TRIAL: NCT07015502
Title: Self-Dehumanization and Hesitation to Report Domestic Violence
Acronym: DESHUMA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A01198-39
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Domestic Violence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Questionnaires
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will undergo socio-demographic and history of violence suffered interview, passation of the Montgomery-Asberg Depression Rating Scale (MADRS),Childhood Trauma Questionnaire, Deshumanization Measure within Romantic Relationships scale, self-esteem scale, violentometer and an implicit association test (IAT).

SUMMARY:
The patients included in the study will be adult women who are victims of domestic violence, consulting for this reason. The duration of participation of each patient will be one hour.

After obtaining the patient's non-opposition to her participation in the study, socio-demographic and history of violence suffered will be collected during an interview with the doctor/nurse. After that, the hetero-questionnaire MADRS (Montgomery-Asberg Depression Rating Scale) will be administered to the patient. This first part will last 30 minutes.

The second part of the study, carried out immediately after the interview, will be carried out on computer in the form of 4 self-questionnaires (Childhood Trauma Questionnaire, Deshumanization Measure within Romantic Relationships scale, self-esteem scale, violentometer) and an implicit association test (IAT). This second part will last 30 minutes.

Then, the participation of the patient in the study is over.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18
* Victim of physical and/or psychological domestic violence taken into care for this reason, following an initial complaint
* Understanding and speaking French
* Subject affiliated to a social security scheme

Exclusion Criteria:

* Patient under legal protection measure (guardianship or legal protection)
* Presence of a disabling mental or cognitive disorder
* Patient employed by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women victims of domestic violence
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Assessment of the correlation between the process of personal dehumanization in victims of domestic violence and their hesitation to file a complaint against the aggressor partner. | 1 year
  To assess the correlation between the process of personal dehumanization in victims of domestic violence and their reluctance to file a complaint against the aggressor partner. This assessment will be based specifically on measuring the time, in number of days, elapsed between the start of the violence and the filing of a complaint.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH Henri Laborit, Poitiers, Vienne (86)
  - CHU Poitiers, Poitiers, Vienne (86)

IPD SHARING:
Plan to Share IPD: No